CLINICAL TRIAL: NCT02341027
Title: Immediate Versus Interval Postpartum Use of the Levonorgestrel Contraceptive Implants: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Mulago Hospital, Uganda (Other); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SFP2016
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Contraceptive Implant Utilization; Lactation
Keywords: Immediate postpartum contraception; Contraceptive implants; Breastfeeding; Jadelle; Lactation; Levonorgestrel
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levonorgestrel (LNG) implants immediately postpartum (Active Comparator): LNG contraceptive implants provided within 5 days of delivery
  Interventions: Device: Jadelle
- Levonorgestrel (LNG) implants 6 weeks postpartum (Active Comparator): LNG contraceptive implants provided 6-8 weeks postpartum
  Interventions: Device: Jadelle

INTERVENTIONS:
Device: Jadelle — within 5 days of delivery and before discharge from hospital
  Other Names: Levonorgestrel contraceptive implants; Sino-Implant
  Arms: Levonorgestrel (LNG) implants immediately postpartum
Device: Jadelle — 6-8 weeks (42-56 days) postpartum
  Other Names: Levonorgestrel contraceptive implants; Sino-Implant
  Arms: Levonorgestrel (LNG) implants 6 weeks postpartum

SUMMARY:
This study will evaluate if immediate postpartum placement of a levonorgestrel (LNG) contraceptive implant within 5 days of delivery improves implant utilization at 6 months postpartum compared to implant placement at 6-8 weeks postpartum among women in Uganda.

DETAILED DESCRIPTION:
Waiting until 6 weeks postpartum to initiate contraception puts women at risk for unintended pregnancy and short birth intervals. Short birth intervals of less than 18 months are associated with an increased risk of preterm delivery and low birth weight infants.

Subdermal implants are advantageous for the postpartum period because they are long-acting, reversible, and highly effective, and they do not contain estrogen or require intrauterine placement. In observational studies postpartum continuation rates have been shown to be greater than 95% after 6 months and 86-87% after 1 year in US populations. Implants are not routinely available during the immediate postpartum period in Uganda, and availability could improve the contraceptive method mix for postpartum women in that country. The results of this study may support increasing access to a form of immediate postpartum LARC (long acting reversible contraception) in a developing country.

This is a randomized, controlled trial of the association between immediate postpartum contraceptive implant placement and implant utilization at 6 months postpartum among women in Uganda. This study will compare the proportion of women using the Levonorgestrel contraceptive implant at 6 months after delivery in women randomized to insertion within 5 days of delivery (immediate insertion) or 6 weeks after delivery (delayed insertion). The study population is women who have a delivery at Mulago hospital in Kampala, Uganda and choose a contraceptive implant for postpartum contraception.

The investigators plan to enroll 202 women who are planning to receive a postpartum Levonorgestrel contraceptive implant after delivery to find out whether the timing of postpartum administration of the implant (prior to hospital discharge or 6 weeks after delivery) affects implant utilization, satisfaction with the implant, vaginal bleeding or breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 - 50 years old
* Voluntarily requesting contraceptive implants for postpartum contraception
* Vaginal delivery or cesarean delivery at Mulago Hospital
* Willing and able to give informed consent
* Agree to a possible home visit for follow up
* Access to a cellphone for the duration of the study

Exclusion Criteria:

* Current breast cancer or breast cancer within the past 5 years
* Decompensated cirrhosis or a liver tumor
* Unexplained vaginal bleeding prior to pregnancy
* Current (or planned) use of Efavirenz medication

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 205 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Implant utilization as measured by the proportion of women using LNG contraceptive implants at 6 months after delivery in women randomized to insertion within 5 days of delivery (immediate insertion) or 6-8 weeks after delivery (delayed insertion). | 6 months

SECONDARY OUTCOMES:
Breastfeeding continuation rates as measured by self-report over the initial 6 months. | 6 months
Time to lactogenesis measured by self-reported onset of lactogenesis. | 72 hours
Change in percentile in infant weight, length and head circumference from delivery to 6 weeks and from delivery to 6 months. | Birth to 6 months
Pregnancy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Averbach, MD, Principal Investigator — University of California, San Francisco; Jody Steinauer, MD, MAS, Principal Investigator — University of California, San Francisco; Josephat Byamugisha, MBChB, PhD, Principal Investigator — Mulago Hospital and Makerere University College of Health Sciences
Locations (1):
- Mulago Hospital, Kampala, Uganda

REFERENCES:
- [Derived] Averbach S, Kakaire O, Kayiga H, Lester F, Sokoloff A, Byamugisha J, Dehlendorf C, Steinauer J. Immediate versus delayed postpartum use of levonorgestrel contraceptive implants: a randomized controlled trial in Uganda. Am J Obstet Gynecol. 2017 Nov;217(5):568.e1-568.e7. doi: 10.1016/j.ajog.2017.06.005. Epub 2017 Jun 10. PMID 28610898